CLINICAL TRIAL: NCT05763290
Title: Childhood Cancer Survivors' Affective Response to Exercise
Status: Recruiting | Type: Observational
Sponsor: St. Jude Children's Research Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: CAREX
Record Dates: First submitted 2023-02-22; First posted 2023-03-10 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: ALL, Childhood; Acute Lymphoblastic Leukemia
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Affective Response to Exercise — Participants will perform a total of three trials of a cognitive task before and after their scheduled SJLIFE cardiovascular stress testing. Participants will then be asked to participate in a qualitative interview about the cognitive task tool and body sensations and emotions experienced during exercise.

SUMMARY:
The primary objective of this study is to assess the feasibility of administering the Personalized Single-Category Implicit Association Test (PSC-IAT) to young adult survivors of childhood cancer.

Participants will perform a total of three trials of a cognitive task before and after their scheduled SJLIFE cardiovascular stress testing. Participants will then be asked to participate in a qualitative interview about the cognitive task tool and body sensations and emotions experienced during exercise.

DETAILED DESCRIPTION:
Researchers at St. Jude Children's Research Hospital want to learn about the measurement of implicit association bias towards or against exercise in childhood cancer survivors. Additionally, researchers want to learn more about the physical and emotional experience of exercise from our survivors.

The plan for this study is to administer single category implicit association tests (PSC-IAT's) to participants during on campus SJLIFE testing and use this data to determine the feasibility of this tool's use in survivors of childhood cancer without cognitive impairment. This study will also administer the Behavioral Regulations in Exercise Questionnaire (BREQ-2)37 to participants as a construct validity check to the PSC-IAT.

The procedures include PSC-IAT and BREQ-2 tests (before and after strenuous exercise as part of the SJLIFE protocol) and a qualitative interview. These will be in addition to standard components of the SJLIFE on-campus visit.

ELIGIBILITY:
Inclusion Criteria:

* Participants enrolled in St. Jude Lifetime Cohort (SJLIFE) aged 18-39 years at completion of on campus visit
* Primary diagnosis of acute lymphoblastic leukemia (ALL)
* No cranial radiation therapy (CRT) as part of treatment for ALL
* Identify as physically inactive (do not meet Centers for Disease Control and Prevention (CDC) guidelines of 150 minutes of moderate physical activity per week or 75 minutes of vigorous physical activity per week)
* Women who are not currently pregnant

Exclusion Criteria:

* Individuals who cannot speak, read, and/or understand English.
* Individuals with an estimated IQ of <70 and/or per PI discretion
* Individuals with any contraindication to stress testing (i.e. cardiovascular complications)
* Women who are currently pregnant

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: The study population will include survivors from the SJLIFE cohort from the ALL diagnostic group (treated without cranial radiation therapy (CRT). This group was chosen because of the prevalence of ALL in childhood cancer diagnoses, and to attempt to prevent potential difficulties with the cognitive task due to cognitive impairment from CRT.
Sampling Method: Non-Probability Sample
Enrollment: 125 (Estimated)
Dates: Start 2023-03-22 (Actual); Primary Completion 2027-02 (Estimated); Study Completion 2030-02 (Estimated)

PRIMARY OUTCOMES:
Implicit Association Bias Testing | Before and after Cardiovascular Stress Testing at Baseline
  Participants' implicit associations with exercise will be measured using the Personalized Single-Category Implicit Association test (PSC-IAT).
Behavioral Regulation of Exercise Questionnaire (BREQ-2): | Before and after Cardiovascular Stress Testing at Baseline
  The Behavioral Regulation of Exercise Questionnaire (BREQ-2) will be administered once to participants in this study to assess trait-level affective motivation.

CONTACTS AND LOCATIONS:
Overall Officials: Megan Ware, MS, PhD, Principal Investigator — St. Jude Children's Research Hospital; Deo Srivastava, PhD, Principal Investigator — St. Jude Children's Research Hospital; Lisa Jacola, PhD, ABPP-CN2, Principal Investigator — St. Jude Children's Research Hospital; Rachel Webster, PhD, Principal Investigator — St. Jude Children's Research Hospital; Tara Brinkman, PhD, Principal Investigator — St. Jude Children's Research Hospital; Kevin Krull, PhD, Principal Investigator — St. Jude Children's Research Hospital; Melissa Hudson, MD, Principal Investigator — St. Jude Children's Research Hospital; Leslie Robinson, PhD, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States